CLINICAL TRIAL: NCT03545958
Title: Exercise to Improve the Hearts and Minds of Canadian Older Adults With Hypertension: The Heart & Mind Study
Brief Title: The Heart & Mind Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Robert Petrella, Associate Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111686
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Hypertension; Cognitive Decline; Vascular Cognitive Impairment
Keywords: Older adults; Community-based; High-intensity interval training (HIT); Mind-motor training
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Research Coordinator will manage recruitment and enrolment of study participants, and will not be involved in either measurement or the intervention. Research personnel performing the outcome assessments and data analysis will be blinded to group allocation but it is not possible to blind participants and personnel delivering the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity Interval Training (HIT) (Experimental): Participants in this groups will receive 15 minutes in the mind-motor training (i.e., Square-Stepping Exercise) followed by a 45-minute HIT intervention.
  Interventions: Behavioral: High-intensity Interval Training (HIT)
- Moderate-intensity Continuous Training (MCT) (Active Comparator): Participants in this groups will receive 15 minutes in the mind-motor training (i.e., Square-Stepping Exercise) followed by a 45-min MCT intervention.
  Interventions: Behavioral: Moderate-intensity Continuous Training (MCT)

INTERVENTIONS:
Behavioral: High-intensity Interval Training (HIT) — Following the mind-motor training component, participants in the experimental group will then continue in the 45-minute HIT intervention, which will be composed by a 10-minute warm-up, a 25-minute core activity, and a 10-minute cool down. The 25-minute core activity will be carried out based on a 4 x 4 minutes aerobic interval training model. The intensity in each cycle will be prescribed at an individual level, and training heart rates will be determined via a sub-maximal excise testing at baseline and monitored during exercise using a wrist-based heart rate monitor (Suunto). In order to ensure progression in aerobic training over the 6-month intervention, training heart rates will be recalculated at the intervention midpoint (i.e., 3 months), where a new sub-maximal exercise test will be performed. Participants will exercise 60 minutes/day, 3 days/week for 6 months.
  Arms: High-intensity Interval Training (HIT)
Behavioral: Moderate-intensity Continuous Training (MCT) — After the mind-motor training component, participants in the comparison/control group will then continue in the 45-min MCT intervention, which will be composed by a 10-minute warm-up a 25-minute moderate-intensity continuous aerobic exercise training, and a 10-minute cool down. The exercise intensity will be prescribed at an individual level, and training heart rates will be determined via a sub-maximal excise testing at baseline and monitored during exercise using a wrist-based heart rate monitor (Suunto). In order to ensure progression in aerobic training over the 6-month intervention, training heart rates will be recalculated at the intervention midpoint (i.e., 3 months), where a new sub-maximal exercise test will be performed. Participants will exercise 60 minutes/day, 3 days/week for 6 months.
  Arms: Moderate-intensity Continuous Training (MCT)

SUMMARY:
Older adults with subjective cognitive decline (SCD) may represent a portion of the population experiencing early sings of cognitive decline. Systolic hypertension is a major contributor to cognitive impairment. High-intensity aerobic interval training (HIT) yields greater fitness and vascular health improvements compared to moderate-intensity aerobic continuous training (MCT). No randomized controlled trials, however, have investigated the effects HIT or MCT on cognition in older adults with hypertension and SCD. Much less is known regarding whether combining HIT or MCT with mind-motor training would culminate additive benefits to cognition. Therefore, the overarching goal of our research is to deliver a group-based exercise program combining mind-motor training with HIT or MCT to older adults with hypertension and SCD. Participants will be randomized into two groups. Participants in both groups will receive 15 minutes of square stepping exercise (SSE) followed by either 45 minutes of HIT (N=70) or 45 minutes of MCT (N=70). In total, both groups will exercise 60 min/day, 3 days/week for 6 months. The effects of both interventions will be evaluated on systolic and diastolic office/ambulatory blood pressure and global and domain-specific cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older;
* Present with controlled or uncontrolled stage 1 hypertension (seated, resting clinic SBP 140 to 179 mmHg and/or DBP 90 to 109 mmHg) as per Hypertension Canada's 2017 Guidelines;
* Have preserved instrumental activities of daily living (scoring >6/8 on the Lawton-Brody Instrumental Activities of Daily Living [IADL] scale);
* Present signs of SCD (defined as answering yes to the question: "Do you feel like your memory or thinking skills have gotten worse recently?");
* Report being concerned about SCD (defined as answering yes to the question: "If yes, are you concerned about the worsening of your memory or thinking skills?");
* Preserved objective cognitive performance (i.e., no signs of MCI or dementia) defined by scoring ≥ 26 on the Montreal Cognitive Assessment (MoCA);
* Must be able to provide written informed consent.

Exclusion Criteria:

* Present signs of objective cognitive impairment (i.e., signs of MCI or dementia), defined by scoring ≤ 25 on the MoCA combined with study physician consult;
* Present resting stage 2 hypertension (seated, resting clinic SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg);
* Present significant neurological conditions or psychiatric disorders (e.g., Parkinson's disease or stroke <1 year); 4) present history of severe cardiovascular conditions (e.g., recent [<1 year] myocardial infarction, left ventricular hypertrophy) and symptomatic cerebrovascular disease;
* Present significant orthopaedic conditions (e.g., severe osteoarthritis in the lower limbs);
* Present untreated clinical depression (i.e., score >15 on the Center for Epidemiologic Studies - Depression scale combined with study physician consult);
* Unable to comprehend the study letter of information. Participants will also be excluded for any other factors that could potentially limit their ability to fully participate in the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Composite score from Cambridge Brain Sciences Cognitive Battery | Change from 0 to 6 months
  Global cognitive functioning assessment
Automated office Systolic Blood Pressure | Change from 0 to 6 months
  Resting blood pressure

SECONDARY OUTCOMES:
24-hour Blood Pressure monitoring | Change from 0 to 6 months
  Ambulatory blood pressure assessment
Maximal oxygen uptake (VO2max) | Change from 0 to 6 months
  Cardiorespiratory fitness assessment
Trail-Making Test | Change from 0 to 6 months
  Executive Functioning assessment
Memory | 0 to 6 months
  Composite measure derived from the Cambridge Brain Sciences cognitive battery (Hampshire, Highfield, Parkin, & Owen, 2012). The composite score is derived from 4 cognitive tasks: Monkey Ladder (visuospatial working memory), Spatial Span (short-term memory), Digit Span (verbal working memory), and Paired Associates (visuospatial learning). For each of the cognitive tasks, higher scores indicate better outcomes. The scores from each task are standardized and averaged to generate a standardized composite measure of memory, i.e., z scores with a mean of 0 and a standard deviation of 1. The standardized scores can range from negative infinity to positive infinity.
Reasoning | 0 to 6 months
  Composite measure from the Cambridge Brain Sciences cognitive battery. The composite score is derived from 3 cognitive tasks: Grammatical Reasoning (verbal reasoning), Double Trouble (modified Stroop task), and Odd One Out (deductive reasoning). For each of the cognitive tasks, higher scores indicate better outcomes. The scores from each task are standardized and averaged to generate a standardized composite measure of reasoning, i.e., z scores with a mean of 0 and a standard deviation of 1. The standardized scores can range from negative infinity to positive infinity.
Planning | 0 to 6 months
  Composite measure from the Cambridge Brain Sciences cognitive battery. The composite score is derived from 2 cognitive tasks: Spatial Planning (planning and executive function) and Token Search (working memory and strategy). For each of the cognitive tasks, higher scores indicate better outcomes. The scores from each task are standardized and averaged to generate a standardized composite measure, i.e., z scores with a mean of 0 and a standard deviation of 1. The standardized scores can range from negative infinity to positive infinity.
Concentration | 0 to 6 months
  Composite measure from the Cambridge Brain Sciences cognitive battery. The composite score is derived from 3 cognitive tasks: Rotations (mental rotation), Feature Match (feature-based attention and concentration), and Polygons (visuospatial processing). For each of the cognitive tasks, higher scores indicate better outcomes. The scores from each task are standardized and averaged to generate a standardized composite measure, i.e., z scores with a mean of 0 and a standard deviation of 1. The standardized scores can range from negative infinity to positive infinity.

OTHER OUTCOMES:
Dual-Task Gait Velocity | 0 to 6 months
  Dual-task velocity is measured in centimetres/second and will be assessed via an electronic walkway (GAITRite® System, 420 cm long, 90 cm wide; CIR Systems). Participants will complete: 1) a single-task walking trial at their own pace; followed by two dual-task walking trials: 2a) walking while naming animals (at baseline) or vegetables (at study endpoint) and 2b) walking while subtracting serial sevens from 90 (at baseline) or 80 (at study endpoint).
Dual-Task Gait Step Length | 0 to 6 months
  Dual-task step length is measured in centimetres and will be assessed via an electronic walkway (GAITRite® System, 420 cm long, 90 cm wide; CIR Systems). Participants will complete: 1) a single-task walking trial at their own pace; followed by two dual-task walking trials: 2a) walking while naming animals (at baseline) or vegetables (at study endpoint) and 2b) walking while subtracting serial sevens from 90 (at baseline) or 80 (at study endpoint).
Dual-Task Gait Variability | 0 to 6 months
  Dual-task gait variability is derived from cycle time variability, measured as the coefficient of variation (%) for cycle time, and will be assessed via an electronic walkway (GAITRite® System, 420 cm long, 90 cm wide; CIR Systems). Participants will complete: 1) a single-task walking trial at their own pace; followed by two dual-task walking trials: 2a) walking while naming animals (at baseline) or vegetables (at study endpoint) and 2b) walking while subtracting serial sevens from 90 (at baseline) or 80 (at study endpoint).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Petrella, MD, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Western University, Western Centre for Public Health and Family Medicine, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boa Sorte Silva NC, Petrella AFM, Christopher N, Marriott CFS, Gill DP, Owen AM, Petrella RJ. The Benefits of High-Intensity Interval Training on Cognition and Blood Pressure in Older Adults With Hypertension and Subjective Cognitive Decline: Results From the Heart & Mind Study. Front Aging Neurosci. 2021 Apr 15;13:643809. doi: 10.3389/fnagi.2021.643809. eCollection 2021. PMID 33935686